CLINICAL TRIAL: NCT06778577
Title: Comparison of the Efficacy of Ultrasound-guided Suprascapular Nerve Pulsed Radiofrequency Neuromodulation and Intra-articular Steroid Injection in Frozen Shoulder Treatment
Brief Title: The Efficacy of Suprascapular Nerve Radiofrequency and Intra-articular Steroid Injection in Frozen Shoulder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Dostalı Alıyev, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: İ7-492-21
Record Dates: First submitted 2024-11-25; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Frozen Shoulder; Radiofrequency Ablation Treatment; Intra-articular Injection
Keywords: frozen shoulder; radiofrequency ablation treatment; intra-articular injection
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones; Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprascapular nerve radiofrequency group (SCNRFT) (Experimental): SCNRFT+intra-articular steroid and local anesthesic injection with physiotherapy. Suprascapular nerve RFT: Ultrasound-guided SCNRFT 42ºC, 360ms.
  Ultrasound-guided intraarticular injection with 40mg triamcinolone+3 cc %0.5 bupivacaine.
  Physiotherapy: The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise. (stretching, mobilization and ROM exercise, and strengthening)
  Interventions: Procedure: suprascapular nerve radiofrequency group (SCNRFT)
- intra-articular corticosteroid injection (IACI) group (Active Comparator): IACI with physiotherapy. Intra-articular steroid+local anesthesic injection: Receive intra-articular corticosteroid injection. Ultrasound-guided IACI with 3c.c. 0.5% bupivacaine and 40mg triamcinolone.
  Physiotherapy: The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise. (stretching, mobilization and ROM exercise, and strengthening)
  Interventions: Other: intra-articular corticosteroid injection (IACI) group

INTERVENTIONS:
Other: intra-articular corticosteroid injection (IACI) group — IACI can provide rapid effect in pain reliving, reducing inflammation and improving ROM that could increase the compliance of exercise therapy.
  Arms: intra-articular corticosteroid injection (IACI) group
Procedure: suprascapular nerve radiofrequency group (SCNRFT) — SCNRFT is a new choice for treatment of frozen shoulder. The suprascapular nerve is the nerve that is most commonly affected in the condition of a frozen shoulder and it is for this reason that the suprascapular nerve is directly targeted by pulsed radiofrequency treatment. As radiology techniques advance, ultrasound-guided SCNB becomes more popular. It provides a cost and time-effective way to "tag" the nerve accurately without injury to the nerves or vessels.
  Arms: suprascapular nerve radiofrequency group (SCNRFT)

SUMMARY:
The aim of this clinical study is to compare the effectiveness of suprascapular nerve pulsed radiofrequency and intra-articular steroid injection in patients with frozen shoulder (adhesive capsulitis). The main questions it aims to answer are:

1. What is the effectiveness of intra-articular steroid injection in frozen shoulder?
2. What is the effectiveness of suprascapular nerve radiofrequency in frozen shoulder?
3. Should these two methods be used together in frozen shoulder?

ELIGIBILITY:
Inclusion Criteria:

* unilateral side involvement.
* ≥50% loss of passive ROM (external rotation or abduction) in the glenohumeral joint comparing to the unaffected side.
* duration of symptoms ≥3 months.
* age≥ 20year old.
* Patients with VAS ≥4 before the procedure

Exclusion Criteria:

* ever received manipulation of the affected shoulder with/without anesthesia. systemic disease, severe degeneration, or trauma involving the shoulder. (ie, rheumatoid arthritis, osteoarthritis, history of injury to the labrum or articular cartilage or malignancies in the shoulder region, etc.)
* neurologic diseases such as stroke or peripheral nerve neuropathy that have already affect the activity of shoulder.
* pain or disorders of the cervical spine, elbow, wrist, or hand.
* a history of drug allergy to local or corticosteroids.
* Pregnancy or lactation.
* Received corticosteroids, or hyaluronic acid intra-articular injection into the affected shoulder during the preceding 4 weeks.
* Patients with VAS <4 before the procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change of The Visual Analogue Scale (VAS) | baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.

SECONDARY OUTCOMES:
The active ROM | Baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The maximal active ROMs of the affected shoulder will be measured using a goniometer under the guidelines of the American Academy of Orthopedic Surgeons. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction.
Change of scores of the Shoulder Pain and Disability Index (SPADI) | Baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Medicine, Department of Anesthesiology and Reanimation, Department of Algology, Ankara, Turkey (Türkiye)